CLINICAL TRIAL: NCT00994071
Title: A Phase I Study of ABT-888, an Oral Inhibitor of Poly(ADP-Ribose) Polymerase and Temozolomide in Children With Recurrent/Refractory CNS Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090243; 09-C-0243
Record Dates: First submitted 2009-10-10; First posted 2009-10-14 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2014-07-16

CONDITIONS: Medulloblastoma; Pontine Glioma; Ependymoma; Astrocytoma; PNET
Keywords: Brain Tumor; CNC Tumor; Pediatric; PARP Inhibitor; Oral Chemotherapy
MeSH Terms: conditions — Medulloblastoma; Ependymoma; Astrocytoma; Neuroectodermal Tumors, Primitive; Brain Neoplasms | interventions — Temozolomide; veliparib

INTERVENTIONS:
Drug: Temozolomide
Drug: ABT-888

SUMMARY:
Background:

- An experimental drug called ABT-888 has been studied in combination with temozolomide (a type of chemotherapy) in adults who have certain kinds of cancer. ABT-88 has been shown to increase tumor sensitivity to temozolomide and improve treatment outcomes in people who have cancer. More research is needed to determine if this combination of drugs will work well as an effective treatment for children who have brain tumors. This will be the first time this combination has been studied in pediatric patients.

Objectives:

* To determine the maximum doses of ABT-888 and temozolomide when given in combination in children with brain tumors.
* To learn how children metabolize and clear ABT-888 from their bodies so that appropriate doses of this medication can be recommended for future clinical trials of this drug.
* To learn what side effects may occur when ABT-888 and temozolomide are given together.
* To learn how certain tumors respond to this combination of drugs by studying the characteristics of these tumors in a laboratory.

Eligibility:

- Individuals less than 21 years of age who have been diagnosed with a cancer of the nervous system (including brain and brain stem tumors) that has not responded to standard therapy.

Design:

* Before beginning the study, participants will have a full medical history and physical examination, and may also be required to have scans of the brain and spine or provide samples of cerebrospinal fluid.
* Treatment will consist of up to 13 28-day cycles of therapy, for a total of 52 weeks (1 year). Participants will receive a dose of ABT-888 twice daily for 5 days, and will receive a dose of temozolomide once daily for 5 days, every 28 days. The morning dose of ABT-888 will be given 60-90 minutes before the dose of temozolomide.
* Participants will have routine blood tests at least once a week throughout the treatment cycles, and will have scans of the brain and spine performed as required by the researchers.

DETAILED DESCRIPTION:
Background

* A subset of patients with pediatric CNS tumors continue to have a poor prognosis despite advances in surgery and radiation. Novel strategies are required for improving outcome for these patients.
* Temozolomide, an oral alkylating agent, has shown modest activity in recurrent pediatric CNS tumors, including high-grade gliomas, medulloblastoma/PNET, and low-grade gliomas.
* Temozolomide induces single-stranded DNA breaks, the majority of which are repaired by the base excision repair (BER) pathway. Poly(ADP-ribose) polymerase, or PARP, is a critical nuclear enzyme that binds to DNA breaks, recruits and activates key proteins in the BER and other DNA repair pathways, halts DNA replication, and facilitates repair of damaged DNA.
* ABT-888 is a potent and orally bioavailable PARP inhibitor that has been shown to enhance cytotoxicity of temozolomide and other chemotherapy agents in several pre-clinical models of human tumors.

Objectives

* To estimate the maximum tolerated dose (MTD) of ABT-888 in combination with temozolomide in children with recurrent or refractory CNS tumors.
* To study the plasma pharmacokinetics (PK) of ABT-888 and PARP inhibition in peripheral blood mononuclear cells (PBMC) in order to recommend a Phase 2 dose of ABT-888 in combination with temozolomide in children with recurrent or refractory CNS tumors.
* To describe the toxicities of the combination of ABT-888 and temozolomide in children with recurrent or refractory CNS tumors.

Eligibility

* Patient must be less than or equal to 21 years of age at registration.
* Patients with a diagnosis of a primary CNS malignancy (including low-grade glioma) that is recurrent or refractory to standard therapy and for which there is no known curative therapy Progression and recurrence will be documented by review of MRI scans. If time permits we will have the diagnosis confirmed by the NCI Laboratory of Pathology. Patients with intrinsic brain stem tumors must have radiographic evidence of progression.
* Karnofsky Performance Scale (KPS for greater than 16 yrs of age) or Lansky Performance Score (LPS for less than or equal to 16 years of age) greater than or equal to 50 assessed within two weeks of study enrollment.
* Patients must have recovered from the toxic effects of all prior therapy.
* Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to registration.

Design

-ABT-888 will be given twice daily on day 1-5, and temozolomide will be given once daily on day 1-5, every 28 days. The morning dose of ABT-888 will be given 60-90 minutes prior to temozolomide.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age:

Patients must be less than or equal to 21 years of age at the time of study enrollment. At the time the MTD or the dose to be recommended for future trials is identified, up to 12 additional patients will be enrolled at that dose level to further define the toxicity profile. Six of these patients will be less than 12 years of age and the other half will be greater than or equal to 12 years.

Tumor:

Patients with a diagnosis of a primary CNS malignancy (including low-grade glioma) that is recurrent or refractory to standard therapy and for which there is no known curative therapy. All patients must have had histological verification of malignancy at initial diagnosis or relapse, excluding patients with diffuse intrinsic brain stem tumors, optic pathway tumors or CNS germ cell tumors with elevations of reliable serum or CSF tumor markers (alpha-fetoprotein or beta-HCG). Patients with intrinsic pontine gliomas or optic pathway tumors do not require histological confirmation of disease but should have clinical and/or radiographic evidence of progression.

Performance Status:

Patients must have Karnofsky Performance Score (for patients greater than 16 years of age) or Lansky Performance Score (for patients less than or equal to 16 years of age) greater than or equal to 50% assessed within two weeks of study enrollment.

Neurological Status:

Patients must be able to take oral medications (either capsules or liquid). Patients with neurologic deficits must have been stable for a minimum of 1 week prior to study entry. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

Prior/Concurrent Therapy:

Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. Recovery is defined as all AE s, attributable to prior therapy, having improved to grade 2 or better or as outlined below.

* Myelosuppressive chemotherapy:

  * Patients must have received their last dose of known myelosuppressive anticancer chemotherapy at least three (3) weeks prior to study registration.
  * Patients must have received their last dose of nitrosourea (including Gliadel) at least six (6) weeks prior to study registration.
* Biologic agent (anti-neoplastic): Patient must have received their last dose of other biologic agent greater than or equal to 7 days prior to study registration.

  --For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
* Monoclonal antibody treatment: Patient must have received their last dose of monoclonal antibody greater than or equal to 4 weeks prior to registration.
* Radiation - Patients who have had prior radiation must have had their last fraction of:

  * Craniospinal irradiation or total body irradiation greater than 3 months prior to registration
  * Local irradiation to the primary tumors or other sites (cumulative dose greater than or equal to 40Gy) greater than 3 months prior to registration
  * Palliative irradiation delivered to symptomatic metastatic sites greater than 4 weeks prior to registration.
* Stem Cell Transplant: Patient must be:

  * greater than or equal to 6 months since allogeneic stem cell transplant prior to registration
  * greater than or equal to 3 months since autologous stem cell transplant prior to registration.
* Corticosteroids: Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to registration.
* Growth factors:

  * Off all colony forming growth factor(s) that support platelet or white blood cell count, number or function for at least 1 week prior to registration (filgrastim, sargramostim, erythropoietin).
  * Off Pegylated G-CSF and/or Erythropoiesis Stimulating Protein for at least 14 days prior to registration.
* Temozolomide: Patients who have received temozolomide previously are eligible for this study if they meet all other inclusion and exclusion criteria.

Organ Function: Documented within 14 days of registration and within 7 days of starting treatment.

* Bone Marrow:

  * Hgb greater than 8 gm/dL (transfusion independent)
  * Platelet count greater than 100,000/mm(3) (transfusion independent)
  * Absolute neutrophil count (ANC) greater than 1,500/mm(3)
* Hepatic:

  * Total Bilirubin (sum of conjugated + unconjugated) less than or equal to 1.5 times institutional upper limit of normal (ULN) for age
  * SGPT (ALT) less than or equal to 2.5 times institutional ULN for age
  * Serum albumin greater than or equal to 2 g/dL
* Renal:

  --Creatinine clearance or radioisotope GFR greater than or equal to 70 ml/min/1.73m(2) or a serum creatinine based on age as follows:
* Age less than 5 (years): a Maximum Serum Creatinine (mg/dL) of 0.8
* Age greater than 5 (years) but less than 10: a Maximum Serum Creatinine (mg/dL) of 1
* Age greater than 10 (years) but less than 15: a Maximum Serum Creatinine (mg/dL) of 1.2
* Age greater than 15 (years): a Maximum Serum Creatinine (mg/dL) of 1.5

Pregnancy or Breast-feeding:

Patients must not be pregnant or breast-feeding. Females of reproductive potential must have a negative serum or urine pregnancy test (within 72 hours prior to enrollment). Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method, which includes abstinence.

Signed informed consent which includes consent to participate in the required pharmacokinetic and pharmacodynamic studies prior to registration.

EXCLUSION CRITERIA:

Concomitant Medications:

Patients receiving any of the following medications are not eligible for study entry:

* Anti-cancer therapy
* Investigational agents

Concurrent Illness:

Patients with any clinically significant, unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that would compromise the patient s ability to tolerate protocol therapy or would likely interfere with the study procedures or results.

Seizures:

Patients with uncontrolled seizures are not eligible for study entry.

Hypertension:

* Patients with inadequately controlled systemic hypertension (SBP and/or DBP greater than 95th percentile for age and height
* Patients with a prior history of hypertensive crisis and/or hypertensive encephalopathy

If a BP measurement prior to registration is greater than 95th percentile for age and height, it must be rechecked and documented to be less than 95th percentile for age and height prior to registration. If a patient falls between the height or weight percentiles, site should average the value as appropriate. For patients greater than or equal to 18 years the normal blood pressure should be less than 140/90 mm of Hg. Patients with hypertension are eligible if their blood pressures become less than 95th percentile for age and height after anti-hypertensive medications.

Prior CNS ischemia and/or infarction:

Patients with documented CNS ischemia and/or infarction, whether symptomatic or discovered incidentally without clinical symptoms, will be excluded from study participation.

Inability to Participate:

Patients with an inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2009-09-22; Study Completion 2013-03-19 (Actual)

PRIMARY OUTCOMES:
To estimate the maximum tolerated dose (MTD) of ABT-888 in combination with Temozolomide in children with recurrent or refractory CNS tumors
-To study the plasma pharmacokinetics (PK) of ABT-888 and PARPinhibition in peripheral blood mononuclear cells (PBMC) in order torecommend a Phase 2 dose of ABT-888 in combination with temozolomide in children with recurrent or refractory ...

SECONDARY OUTCOMES:
To measure non-homologous end-joining (NHEJ) activity in peripheral blood mononuclear cells (PBMC) prior to and following ABT-888 administration.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Warren, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Newlands ES, Stevens MF, Wedge SR, Wheelhouse RT, Brock C. Temozolomide: a review of its discovery, chemical properties, pre-clinical development and clinical trials. Cancer Treat Rev. 1997 Jan;23(1):35-61. doi: 10.1016/s0305-7372(97)90019-0. No abstract available. PMID 9189180
- [Background] Sankar A, Thomas DG, Darling JL. Sensitivity of short-term cultures derived from human malignant glioma to the anti-cancer drug temozolomide. Anticancer Drugs. 1999 Feb;10(2):179-85. doi: 10.1097/00001813-199902000-00006. PMID 10211548
- [Background] Patel M, McCully C, Godwin K, Balis FM. Plasma and cerebrospinal fluid pharmacokinetics of intravenous temozolomide in non-human primates. J Neurooncol. 2003 Feb;61(3):203-7. doi: 10.1023/a:1022592913323. PMID 12675312